CLINICAL TRIAL: NCT06782529
Title: Comparison of Varying Doses of Steroid for Intra-articular Knee Injections
Brief Title: Knee Injections for Obese Patients With Knee Arthritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jeff P. Nadwodny, Assistant Professor of Family Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-005200
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis of Knee
Keywords: Knee Osteoarthritis; Corticosteroid Injection; Obesity
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Dose Group (Active Comparator): Patients with knee osteoarthritis who are interested in knee intra-articular corticosteroid injections and meet the inclusion criteria.
  Interventions: Drug: Triamcinolone Acetonide Standard Dose
- Lower Dose Group (Experimental): Patients with knee osteoarthritis who are interested in knee intra-articular corticosteroid injections and meet the inclusion criteria.
  Interventions: Drug: Triamcinolone Acetonide Low Dose

INTERVENTIONS:
Drug: Triamcinolone Acetonide Low Dose — Subjects will receive a reduced dose of 20mg of triamcinolone acetonide.
  Total injection volume of 5ml, consisting of:
  * 0.5ml triamcinolone acetonide (20mg)
  * 4.5ml lidocaine (45mg)
  Arms: Lower Dose Group
Drug: Triamcinolone Acetonide Standard Dose — Subjects will receive the standard of care dose of 40mg triamcinolone acetonide
  Total injection volume of 5ml, consisting of:
  * 1ml triamcinolone acetonide (40mg)
  * 4ml lidocaine (40mg)
  Arms: Standard Dose Group

SUMMARY:
The purpose of this study is to assess obese patients with knee arthritis and determine the non-inferiority of a low dose steroid treatment vs. standard dose steroid treatment for two knee outcome measures: pain and function.

ELIGIBILITY:
Inclusion Criteria:

• Patients with BMI ≥30 kg/m2 and radiograph-proven knee osteoarthritis who are interested in receiving a steroid injection for knee arthritis.

Exclusion Criteria:

* BMI < 30 kg/m2
* Uncontrolled diabetics with a hemoglobin A1c > 8%
* No other treatment within the time frame of the study.
* Patients that are undergoing physical therapy at the time of the study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-01-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Scale (NPS) | Baseline, 4 weeks, 12 weeks
  The Numerical Pain Scale (NPS) uses a 0-10 point rating system in which the patient selects the number that describes their current pain level, where "0" represents "no pain" and "10" represents "the worst pain imaginable"
Knee Injury and Osteoarthritis Outcome score (KOOS) | Baseline, 4 weeks, 12 weeks
  The Knee Injury and Osteoarthritis Outcome is a commonly used questionnaire which focuses on how patients are affected by osteoarthritis symptoms in five areas: knee pain, stiffness, daily activity, sport and recreation, and quality of life. Results are scored 0-100. 0 = extreme problems, 100 = no problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey P Nadwodny, DO, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials